CLINICAL TRIAL: NCT04597359
Title: A Phase II Randomized Double Blinded Study of Green Tea Catechins (GTC) vs. Placebo in Men on Active Surveillance for Prostate Cancer: Modulation of Biological and Clinical Intermediate Biomarkers
Brief Title: To Evaluate if Green Tea Can be Effective in Reducing the Progression of Prostate Cancer in Men on Close Monitoring
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EA8184; NCI-2020-07173 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA8184 (Other: ECOG-ACRIN Cancer Research Group); ECOG-ACRIN-EA8184 (Other: DCP); EA8184 (Other: CTEP); UG1CA189828 (NIH)
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — green tea extract polyphenone E; polyphenon E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (green tea catechins) (Experimental): Patients receive green tea catechins PO BID for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Sinecatechins
- Arm B (placebo) (Placebo Comparator): Patients receive placebo PO BID for up to 6 months.
  Interventions: Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Placebo Administration — Given PO
  Arms: Arm B (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Sinecatechins — Given PO
  Other Names: Camellia sinensis Leaf Catechins; Kunecatechins; Polyphenon E; Polyphenon E TM; Veregen
  Arms: Arm A (green tea catechins)

SUMMARY:
This phase II trial studies how well green tea catechins work in preventing progression of prostate cancer from a low risk stage to higher risk stages in men who are on active surveillance. Green tea catechins may stabilize prostate cancer and lower the chance of prostate growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the change in the percent (%) Ki-67 expression in a biopsy core positive for cancer from baseline to end-of-study (EOS) biopsy between men on active surveillance (AS) for prostate cancer (PCa), treated with green tea catechins (GTCs) or placebo for 6 months.

SECONDARY OBJECTIVES:

I. To assess apoptosis by caspase in tumor tissue from EOS biopsy by treatment. II. To assess % Ki-67: Apoptosis ratio from EOS biopsy by treatment. III. To evaluate the number of biopsy cores positive for cancer from EOS biopsy by treatment.

IV. To evaluate the percentage of any biopsy tissue core positive for cancer from EOS biopsy by treatment.

V. To evaluate % Ki-67 in EOS biopsy from the same quadrant matching the quadrant with the highest % Ki-67 at baseline treatment.

VI. To evaluate the Gleason sum from EOS biopsy by treatment. VII. To evaluate the change in serum prostate-specific antigen (PSA) from baseline to 3 months and to EOS by treatment.

VIII. To evaluate the safety of 6 month administration of GTC assessed by Common Toxicity Criteria (CTC) version 5.0, complete blood count (CBC), comprehensive metabolic panel (CMP) and liver function toxicities (LFTs) by treatment.

IX. To evaluate the change in geometric mean of % Ki-67 measures in all the cores positive for cancer from baseline to EOS biopsy by treatment.

EXPLORATORY OBJECTIVES:

I. To evaluate the change in catechin (epigallocatechin gallate [EGCG]) as indicated by change from EGCG measured in plasma from baseline and EOS by treatment.

II. To evaluate the adherence and acceptability to GTC based on the percentage compliance using agent logs (%) and pill counts monthly until EOS by treatment groups.

III. To evaluate the bioavailability of GTC as indicated by change from EGCG measured in plasma from baseline and EOS by treatment groups.

PATIENT REPORTED OUTCOMES OBJECTIVES:

I. To evaluate the change in lower urinary tract symptoms (LUTS) from baseline to 3 months and to EOS using the LUTS scale by treatment groups.

II. To evaluate the change in quality of life (QOL) scores from baseline to 3 months and to EOS using the Functional Assessment of Cancer Therapy (FACT)-Prostate by treatment groups.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive green tea catechins orally (PO) twice daily (BID) for up to 6 months in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive placebo PO BID for up to 6 months.

After completion of study, patients are followed up at approximately 7 days, at 6 months, and then up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA FOR PREREGISTRATION (STEP 0: SCREENING)
* Patient must have biopsy-proven (consisting of >= 12 tissue cores) adenocarcinoma of the prostate with cancer present in at least one biopsy core in the most recent biopsy using initial transrectal ultrasound (TRUS) biopsy or TRUS biopsy followed by multiparametric magnetic resonance imaging (mpMRI) of the prostate and a confirmatory targeted biopsy
* Patient must be on active surveillance (very low, low and favorable intermediate risk as defined by the National Comprehensive Cancer Network [NCCN])
* Patient must be scheduled for a follow up prostate biopsy 6 months after the initiation of treatment on this study
* Patient must have a serum PSA < 10 ng/mL or prostate specific antigen density (PSAD) < 0.15 ng/mL/ g obtained within 30 days of registration
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patient must be willing to abstain from consumption of any supplements containing green tea catechins
* Patient must be willing to restrict tea consumption to less than three (3) servings of hot tea or three (3) servings of iced tea per week (serving size of 8 oz)
* Patient must be willing to discontinue current vitamin/mineral supplement use and use one provided by study
* Patient must be willing to take study agent or placebo at the dose specified with meals
* Patient must have the ability to understand and the willingness to sign a written informed consent document
* Absolute neutrophil count >= 1,200/mm^3 (>= 1.2 k/uL) (obtained within 30 days prior to registration)
* Platelets >= 75,000/mm^3 (>= 75 k/uL) (obtained within 30 days prior to registration)
* Total bilirubin =< 1.2 mg/dL (or =< 3.0 mg/dL for patients with Gilbert's syndrome) (obtained within 30 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x upper limit of normal (ULN) (obtained within 30 days prior to registration)
* Serum creatinine =< 1.5 x ULN (obtained within 30 days prior to registration)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Sexually active males must use an accepted and effective method of double barrier contraception (vasectomy must be combined with a physical barrier method) or abstain from sexual intercourse for the duration of their participation in the study
* Patients must have archived formalin-fixed paraffin-embedded (FFPE) tumor tissue specimen available for Gleason score confirmation and % Ki-67 expression (5% or more) in tumor tissue for eligibility and stratification. Tumor tissue can be submitted any time during screening

  * Tumor tissue specimen has been collected and is ready to ship to H. Lee Moffitt Cancer Center & Research Institute

    * H. Lee Moffitt Cancer Center & Research Institute will perform Gleason score confirmation and % Ki-67 expression (5% or more) in tumor tissue and notify the Eastern Cooperative Oncology Group-American College of Radiology Imaging Network (ECOG-ACRIN) Operations Office and submitting institution within 3-4 business days of receipt of the tumor tissue specimen
* INCLUSION CRITERIA FOR RANDOMIZATION (STEP 1)
* Patient must meet all Step 0 eligibility criteria at the time of their registration to Step 1
* Patient must have Gleason score (3+3) or predominant Gleason pattern 3 (3+4), =< 33% of biopsy cores, and =< 50% involvement of any biopsy core
* Patient must have % Ki-67 expression of 5% or more in tumor tissue

Exclusion Criteria:

* EXCLUSION CRITERIA FOR PREREGISTRATION (STEP 0: SCREENING)
* Patient must not have had prior treatment for prostate cancer, including focal therapy, with surgery, irradiation, local ablative (i.e., cryosurgery or high-intensity focused ultrasound), or androgen deprivation therapy
* Patient must not have a history of renal or hepatic disease, including history of hepatitis B and C
* Patient must not have prostate cancer with distant metastases
* Patient must not have undergone treatment of hormone therapy, immunotherapy, chemotherapy and/or radiation for any malignancies within the past 2 years. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patient must not receive any other investigational agents while on this study
* Patient must not have a history of allergic reactions attributed to tea or other compounds of similar chemical or biologic composition to green tea extracts

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the highest percent Ki-67 expression | Baseline to 6 months
  Measured in a core positive for tumor from baseline to highest percent (%) Ki-67 expression measured in a core positive for tumor in the end of study (EOS) biopsy. This change will be compared between green tea catechins (GTC) and placebo arms. The highest % Ki-67 expressions from baseline and EOS biopsies will be used to estimate the change. If the change is not normally distributed, non-parametric test such as Wilcoxon-rank sum test or two-sample normal score test will be used to compare the changes in percent Ki-67 levels between the GTC and placebo arms.

SECONDARY OUTCOMES:
Apoptosis | Up to 6 months
  Will be assessed by caspase in tumor tissue from EOS biopsy by treatment.
Apoptosis ratio | Up to 6 months
  Will be evaluated from EOS biopsy by treatment groups. Descriptive statistics with confidence intervals will be presented. For continuous measures, will use two-sample t-test or Wilcoxon rank sum test (if non-parametric test is more appropriate) to compare the measurements by treatment.
Number of biopsy cores positive for cancer at end of study | At 6 months
  Descriptive statistics with confidence intervals will be presented. For binary measures, will use Fisher's test.
Percent of any biopsy tissue core positive for cancer at end of study | At 6 months
  Descriptive statistics with confidence intervals will be presented. For continuous measures, will use two-sample t-test or Wilcoxon rank sum test (if non-parametric test is more appropriate) to compare the measurements by treatment.
Percent Ki-67 | Up to 6 months
  Descriptive statistics with confidence intervals will be presented. For continuous measures, will use two-sample t-test or Wilcoxon rank sum test (if non-parametric test is more appropriate) to compare the measurements by treatment.
Gleason sum at end of study | At 6 months
  Descriptive statistics with confidence intervals will be presented. For binary measures, will use Fisher's test.
Change in serum prostate-specific antigen (PSA) | Baseline up to 6 months
  Will use three mixed models (for PSA, PSA doubling time, and PSA density). For the first two, will log the PSA value. For PSA, will have intercepts and slopes for each patient, an unstructured covariance model, and 2 terms for the intercept and slope associated with the treatment group. For the PSA doubling time, will center the baseline values at 1, and estimate the slopes for each patient (from which the doubling time can be derived), along with a net slope effect for the treatment group. The mixed model for PSA density will be analogous to the one for PSA.
Incidence of adverse events | Up to 12 months
  Will be assessed by Common Toxicity Criteria version 5.0, complete blood count, comprehensive metabolic panel, and liver function toxicities by treatment. All toxicity data will be summarized by category and grade in a standard fashion. Proportions experiencing the most common types of toxicity in this trial will be estimated and 95% confidence intervals calculated. Adverse event rates (such as worst grade 3 or higher) by arm will be estimated and compared.
Change in geometric mean of percent Ki-67 | Baseline up to 6 months
  Descriptive statistics with confidence intervals will be presented. For binary measures, will use Fisher's test.

OTHER OUTCOMES:
Compliance to study drug (standard pill counts) | Up to 6 months
  Compliance to study drug will be evaluated by standard pill counts. Will evaluate percentage compliance to study agent in the study arms using pill counts.
Compliance to study drug (diet records) | Up to 6 months
  Compliance to study drug will be evaluated by diet records.
Compliance to study drug (plasma concentrations of GTC) | Up to 6 months
  Compliance to study drug will be evaluated by plasma concentrations of GTC (epigallocatechin gallate [EGCG]). For plasma, will assess the change from baseline to end of treatment for GTC (EGCG) to estimate compliance and bioavailability.
Epigallocatechin gallate (EGCG) concentrations | Up to 6 months
  Will correlate EGCG concentrations with prostate specific antigen density (PSAD) and prostate specific antigen doubling time (PSADT), using descriptive analysis with scatter plots and regression analysis, and adjusting intervention and known predictors including the stratification factors in multivariable analysis. Will transform to the square root or logarithmic transformation of the data to improve normality of the distributions (determined as the transformation (including untransformed) with the lowest Anderson-Darling normality score).
Changes in lower urinary tract symptoms (LUTS) | Baseline up to 6 months
  Lower urinary tract symptoms (LUTS) will be assessed using the American Urological Association Symptom Score for the evaluation, LUTS Symptom Scale. The highest score on the scale is 5, "almost always" and the lowest score on the scale is 0, "not at all".
Changes in lower urinary tract symptoms | Baseline up to 6 months
  Will assess change in EGCG from baseline to EOS, adherence to GTC, and bioavailability of GTC from baseline to EOS by treatment.
Changes in quality of life (QOL) | Baseline up to 6 months
  Quality of life will be assessed using the Functional Assessment of Cancer Therapy (FACT)-Prostate.
Changes in quality of life (QOL) | Baseline up to 6 months
  Will assess change in EGCG from baseline to EOS, adherence to GTC, and bioavailability of GTC from baseline to EOS by treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nagi B Kumar, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (353):
- United States (345):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Marshall Cancer Center, Cameron Park, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Epic Care-Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Mercy Cancer Center, Merced, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Marshall Hospital, Placerville, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - UCSF Cancer Center - San Mateo, San Mateo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - BASS Medical Group - Lennon, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - UCHealth - Cherry Creek, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Straub Pearlridge Clinic, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Mercy Health - Paducah Medical Oncology and Hematology, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Maine Medical Partners Urology, South Portland, Maine
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Hospital Center, Jamaica, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Outer Banks Hospital, Nags Head, North Carolina
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Chesapeake Regional Medical Center, Chesapeake, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
- FHP Health Center-Guam, Tamuning, Guam
- Puerto Rico (7):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan